CLINICAL TRIAL: NCT01108159
Title: Integrated Whole-Genome Analysis of Hematologic Disorders Using High-Throughput Sequencing and Array Technologies
Brief Title: Integrated Whole-Genome Analysis of Hematologic Disorders
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jason D. Merker, Assistant Professor of Pathology, Stanford University
Other Study IDs: HEM0013; 1081737-100-DHAAT; SU-09092009-3820 (Other: Stanford University); 16329 (Other: Stanford IRB)
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Hematologic Diseases
MeSH Terms: conditions — Hematologic Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, bone marrow, skin biopsy

INTERVENTIONS:
Procedure: Blood Draw
Procedure: Skin Biopsy

SUMMARY:
We will use new technologies to look at the DNA, RNA, proteins, and metabolites in the disease-containing blood, bone marrow, or tissue and normal cells from the skin. Our goal is to analyze all of the genes in the diseased and normal skin sample. By comparing the results of the diseased sample and normal skin cells and the results of the two types of genetic information (DNA and RNA), we should be able to identify genetic changes that are important for the initiation, progression, or treatment response of that particular disorder.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Patient meets the clinical and/or pathologic criteria for the hematologic disorder being examined.
3. Patient is willing to provide a skin biopsy and five 10 mL tubes of peripheral blood.

Exclusion Criteria:

1. Less than 18 years of age
2. Patient is not willing to provide a skin biopsy and five 10 mL tubes of peripheral blood.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participants with hematologic disorders
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2009-09; Primary Completion 2013-08-02 (Actual); Study Completion 2013-08-02 (Actual)

PRIMARY OUTCOMES:
to identify mutations, changes in DNA copy number, structural rearrangements, or altered coding and non-coding RNA expression | sample collection at time of routine visit

CONTACTS AND LOCATIONS:
Overall Officials: James L Zehnder, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Merker JD, Roskin KM, Ng D, Pan C, Fisk DG, King JJ, Hoh R, Stadler M, Okumoto LM, Abidi P, Hewitt R, Jones CD, Gojenola L, Clark MJ, Zhang B, Cherry AM, George TI, Snyder M, Boyd SD, Zehnder JL, Fire AZ, Gotlib J. Comprehensive whole-genome sequencing of an early-stage primary myelofibrosis patient defines low mutational burden and non-recurrent candidate genes. Haematologica. 2013 Nov;98(11):1689-96. doi: 10.3324/haematol.2013.092379. Epub 2013 Jul 19. PMID 23872309